CLINICAL TRIAL: NCT00234468
Title: A Phase III, Double-Blind, Randomised Study Comparing ZD1839 (IressaTM) Versus Placebo As Maintenance Therapy In Subjects With Locally Advanced Stage III Non-Small Cell Lung Cancer (NSCLC) After Combined Modality Therapy
Brief Title: Iressa vs Placebo as Maintenance Therapy in Locally Advanced NSCLC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed due to insufficient recruitment
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839IL/0126
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Locally Advanced Non Small Cell Lung Cancer (Stage IIIA and IIIB)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

INTERVENTIONS:
Drug: Iressa (Gefitinib)

SUMMARY:
The aim of the study if to determine if Iressa can prolong the period of time without any disease worsening (Time to progression) in patients previously treated with combined therapy such as surgery and chemotherapy with or without radiotherapy or chemotherapy and radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Histologically Confirmed Non Small Cell Lung Cancer.
* Locally advanced disease previously treated with combined therapy (chemotherapy and surgery with or without radiotherapy, or chemotherapy and radiotherapy).
* Chemotherapy with regimens containing cisplatin or carboplatin is mandatory
* Response to combined therapy

Exclusion Criteria:

* No previous treatment with ZD1839 or any other EGFR-targeted therapy
* No progressive disease after combined therapy for locally advanced NSCLC
* No presence of metastatic disease
* No other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Any unresolved chronic toxicity from previous anticancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2004-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to progression (2 years after Last patient in)

SECONDARY OUTCOMES:
Modalities of relapse or progression (2 years after Last patient in)
Overall survival (2 years after Last patient in)

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Crino, MD, Principal Investigator — Bologna Italy
Locations (32):
- Italy (32):
  - Research Site, Avellino
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Cagliari
  - Research Site, Campobasso
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Chieti
  - Research Site, Cosenza
  - Research Site, Della Fratte
  - Research Site, Emilia
  - Research Site, Fano
  - Research Site, Florence
  - Research Site, Forlì
  - Research Site, Frattamaggiore
  - Research Site, Livorno
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Potenza
  - Research Site, Ravenna
  - Research Site, Rimini
  - Research Site, Roma
  - Research Site, San Giovanni Rotondo
  - Research Site, Sassari
  - Research Site, Taormina
  - Research Site, Venezia-Mestre